CLINICAL TRIAL: NCT02697110
Title: Family Inclusive Early Brain Stimulation
Acronym: FINEBRAINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ibadan (Other)
Collaborators: Grand Challenges Canada (Other)
Responsible Party: Principal Investigator, Dr. A.O. Adebiyi, Coordinator, College of Medicine Research and innovation Management Unit, University of Ibadan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AD/13/479/741
Record Dates: First submitted 2016-02-22; First posted 2016-03-03 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Brain Stimulation
Keywords: Cognition; Brain Stimulation; Early Child Development

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Edutainment based intervention (Experimental): This group receives the usual routine immunization at 6, 10, 14 weeks and 9 months and an Edutainment intervention package of limited group (i.e., 3-5 women) drama based video session (Edutainment) followed by a Question and Answer session with mothers on early brain development, parenting skills, communication and negotiating skills at 6 weeks. Mothers will be encouraged to train fathers and other caregivers at home with reinforcement of key messages at subsequent clinic visits. Key messages will be delivered through the use of flip charts at 14 weeks and given to mothers as take home for use in engaging the fathers partners and other caregivers for their child. Reinforcement of key messages at subsequent visits will be through the use of videos and flip chart.
  Interventions: Behavioral: Edutainment based intervention
- B (No Intervention): This group receives routine immunization care (usually includes group health talk) at 6, 10, 14 weeks and 9 months.

INTERVENTIONS:
Behavioral: Edutainment based intervention — Edutainment intervention package
  Arms: A: Edutainment based intervention

SUMMARY:
Social interaction (in the form of serve and return exchanges) between child and parent are crucial for psychosocial, physical and cognitive development. Parents in sub-Saharan countries are ill-equipped to maximize the benefits from this interaction. The investigators approach builds on the traditional outlook that "it takes a village to raise a child" i.e., not only the parents but other extended family members play a role as caregivers to young children. The investigators intention is to use the existing post-natal/child welfare clinics to deliver an intervention, which uses culturally acceptable videos and active skills building, to deliver health messages and practical skills to women, with the intention that they will subsequently engage and teach their partners and other caregivers about early brain stimulation and child development.

DETAILED DESCRIPTION:
A two arm cluster randomized control design will be used to select a total of about 400 participants each of the control and intervention groups. The participants will be drawn from primary health care (PHC) centres offering immunization services in Ibadan. In the intervention group, mothers will be trained on early brain stimulation using group video sessions followed by individualised question and answer sessions. These sessions will take place at 6 week and 10 week post natal immunisation visits. The control arm will receive the standard of care - routine immunization care- group health talks.

The child's development will be assessed using the Survey of Wellbeing of Young Children (SWYC) instrument.

Outcome variables will include changes in self-reported early child brain stimulation behaviour and increase in the awareness of parents and significant others on the social and emotional difficulties of children.

ELIGIBILITY:
Inclusion Criteria:

* All mothers with live children aged 1-6 weeks

Exclusion Criteria:

* Mothers of children with moderate to severe birth asphyxia or gross congenital anomalies
* Mothers who are unable to communicate to provide information

Ages: 1 Week to 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Actual)
Dates: Start 2014-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Reduction in socio-cognitive deficit as measured by the Survey of Well being of Young Children (SWYC) | 6weeks, 14 weeks, 9months, 12 months and 18 months
  Reduced socio-cognitive deficit in the intervention compared to the control group at 18 months of age
Improved child stimulation practices as measured by assessment of study constructed self-reported child stimulation practices questionnaire | 18 months
  Improved child stimulation practices in the intervention compared to the control group at 18 months of age
Number of children with developmental delays as measured by The WHO head circumference growth curves and WHO Child Growth Standards | 6weeks to 18 months
  Appropriate for Age physical development of children such as Head circumference, Length/height, Weight for Age as measured by The WHO head circumference growth curves and WHO Child Growth Standards

SECONDARY OUTCOMES:
Increased mothers knowledge and competence on child brain stimulation practices as measured by a study constructed domain based questionnaire on knowledge and competence instrument | 9mths -12 months
  An increase in mothers knowledge and competence on child brain stimulation practices
Mothers engagement of fathers and other caregivers on early brain stimulation as measured by simple questionnaire on mothers self-reported father engagement activity | 6-18months
  Mothers are expected to effectively engage their male partners and other caregivers on child development. This will be demonstrated by their success at getting their male partner and other caregivers trained at home.
fathers' self- reported engagement and investment in the early childhood development as measured by study derived adaptations of the "Self-Perceptions of the Parental Role scale (SPPR)" and the Early Childhood Study Survey Tool | 18 months
  fathers' self- reported engagement and investment in the early childhood development would improve (responsible behaviour, emotional engagement, physical accessibility, material support, involvement in child care, influence in child rearing decisions)
Increased knowledge and competence of health workers on early brain stimulation as measured by study derived composite questionnaire on knowledge and competence on intervention | 14weeks - 9months
  The competence and knowledge of health workers to successfully deliver intervention this intervention after being trained would also be a secondary measure of success.

CONTACTS AND LOCATIONS:
Overall Officials: Akindele O Adebiyi, MBchB, MPH, Principal Investigator — College of Medicine University of Ibadan

IPD SHARING:
Plan to Share IPD: Undecided
Decision would be based on research teams final decision after the crucial manuscripts have been published